CLINICAL TRIAL: NCT02711514
Title: Femoral Artery Crossover Rates of 1000 Consecutive Radial (or Ulnar) Artery Procedures in the Cardiac Cath Lab for Diagnostic Cardiac Catheterizations and/or Percutaneous Coronary Interventions
Brief Title: Femoral Artery Crossover Rates in 1000 Consecutive Radial Cath Labs Procedures.
Acronym: FACR
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Miami Cardiac and Vascular Institute (Other)
Responsible Party: Principal Investigator, Raul Herrera, MD, Director Cardiac and Vascular Institute, Miami Cardiac and Vascular Institute
Other Study IDs: JR1000R
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Retrospective Review

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Comparison of Crossover rates of Radial Cardiac Catheterizations and/or PCIs into femoral vs published literature

DETAILED DESCRIPTION:
A retrospective review of 1000 consecutive Radial or Ulnar Cardiac Catheterizations and/or Percutaneous Coronary Interventions performed in our Institute by one single operator could provide us with the cross over rates to femoral interventions. In this manner these rates could be compared to the published rates of other institutions benchmarking our techniques with the outcomes for such interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming to the emergency room requiring Diagnostic Cardiac Catheterizations and/or Percutaneous Coronary Interventions

Exclusion Criteria:

* Cardiac Tamponade
* Cardiogenic Shock

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 Consecutive Patients who underwent Radial (or Ulnar) Artery Procedures in the Cardiac Cath Lab for Diagnostic Cardiac Catheterizations and/or Percutaneous Coronary Interventions.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Crossover rate from Radial to Femoral access | 1 year
  How often do you start a Cath on the Radial Artery and for any reason, have to switch to Femoral Artery.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Quesada, MD, Principal Investigator — Director Structural Heart BHSF
Locations (1):
- Miami Cardiac and Vascular Institute, Miami, Florida, United States